CLINICAL TRIAL: NCT07068542
Title: the Safety and Efficacy of Sacituzumab Tirumotecan Combined With Immunotherapy in Advanced Thyroid Cancer: A Single-arm, Multi-center, Open-label Clinical Study
Brief Title: Sacituzumab Tirumotecan Combined With Immunotherapy in Advanced Thyroid Cancer
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Zhejiang Provincial People's Hospital (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: KY2025070
Record Dates: First submitted 2025-05-14; First posted 2025-07-16 (Actual); Last update posted 2025-07-16 (Actual); Status verified 2025-05

CONDITIONS: Advanced Thyroid Carcinoma; Radioiodine-refractory Differentiated Thyroid Cancer
Keywords: radioiodine-refractory differentiated thyroid cancer; Sacituzumab tirumotecan; immunotherapy; TROP2; anaplastic thyroid carcinoma
MeSH Terms: conditions — Thyroid Carcinoma, Anaplastic | interventions — tislelizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- cohort A (Experimental): Unresectable, locally advanced or metastatic advanced thyroid carcinoma (ATC) will receive Sacituzumab tirumotecan combined with Tislelizumab
  Interventions: Drug: Sacituzumab tirumotecan; Drug: Tislelizumab
- cohort B (Experimental): Unresectable, locally advanced or metastatic radioiodine-refractory differentiated thyroid carcinoma (RAIR-DTC) will receive Sacituzumab tirumotecan combined with Tislelizumab
  Interventions: Drug: Sacituzumab tirumotecan; Drug: Tislelizumab

INTERVENTIONS:
Drug: Sacituzumab tirumotecan — Sacituzumab tirumotecan: 4mg/kg, IV, Q6W, D1, D15, D22
Drug: Tislelizumab — Tislelizumab: 400mg, IV, Q6W, D1

SUMMARY:
This study is a multi-center, phase II clinical trial, primarily enrolling patients with unresectable, locally advanced or metastatic undifferentiated thyroid cancer (ATC) or radioiodine-refractory differentiated thyroid cancer (RAIR-DTC). Eligible patients will receive treatment with Sacituzumab tirumotecan combined with tislelizumab until disease progression or intolerability occurs. The effectiveness and safety will be evaluated.

ELIGIBILITY:
Inclusion Criteria:

1. age ≥18 years
2. Histologically confirmed unresectable or metastatic undifferentiated thyroid carcinoma (ATC), and patients who are unwilling to undergo surgery are also eligible. Histologically confirmed unresectable or metastatic differentiated thyroid carcinoma (DTC), including papillary thyroid carcinoma, follicular thyroid carcinoma (high cell type, thyroid island type, follicular subtype, poorly differentiated thyroid carcinoma or any combination of the above histological types); a) For the ATC cohort: not carrying the BRAF V600E mutation, or carrying the BRAF V600E mutation but having failed previous BRAF-targeted therapy, or carrying the BRAF V600E mutation but refusing BRAF-targeted therapy; b) For the DTC cohort: must be refractory to radioactive iodine (RAI) treatment (i.e., no response to RAI treatment), and the determination criteria are as follows: (a)measurable lesion(s) without radioactive iodine uptake, (b) measurable lesion(s) progressive by RECIST 1.1 and/or the appearance of new lesion(s) within 12 months of prior radioactive iodine therapy, (c) cumulative radioactive iodine dose of >600 mci, or (d) measurable disease that was Fludeoxyglucose (18F) positron emission tomography scan positive.
3. Patients with PDTC must have at least one target lesion by RECIST v1.1.
4. No active autoimmune disease;
5. No concurrent malignant tumors;
6. Expected survival ≥ 12 weeks
7. Lymphocyte count ≥ 1.2 × 10^9/L, Platelet count ≥ 100 × 10^9/L, Hemoglobin ≥ 9.0 g/L
8. AST and ALT ≤ 2.5 × ULN, Total bilirubin ≤ 1.5 × ULN,for patients with documented liver, AST and ALT ≤ 5 × ULN
9. creatinine clearance (CrCl) ≥ 60 mL/min

Exclusion Criteria:

1. Received prior treatment with a trophoblast cell-surface antigen 2 (TROP2)-directed antibody drug conjugate (ADC) or a topoisomerase I inhibitor-containing ADC. Received prior therapy with an agent directed to another stimulatory or coinhibitory T-cell receptor (eg, cytotoxic T-lymphocyte-associated protein-4 [CTLA-4], OX-40 [cluster of differentiation (CD) 134], or CD137)
2. Has known additional malignancy that is progressing or has required active treatment within the past 3 years (Except for those tumors that have been cured by local treatment, such as basal cell carcinoma of the skin, squamous cell carcinoma of the skin, and carcinoma in situ of the cervix, etc.)
3. For presence of brain metastases, if the CNS disease is stable for at least 4 weeks before the first administration and the use of corticosteroids for brain metastases has been stopped for at least 2 weeks before study, they are eligible for inclusion. For subjects with asymptomatic brain metastases without previous treatment are also eligible.
4. Patients experienced myocardial infarction, unstable angina pectoris, acute or persistent myocardial ischemia, grade 3 or 4 heart failure, symptomatic or poorly controlled severe arrhythmia, cerebrovascular accident, transient ischemic attack and other serious cardiovascular and cerebrovascular diseases; has a history of myocardial diseases such as myocarditis, primary cardiomyopathy, or specific cardiomyopathy; any deep vein thrombosis within 3 months prior to administration (if treated with low molecular weight heparin or similar efficacy drugs for ≥ 2 weeks and stabilized, inclusion is allowed); has had peripheral arterial thromboembolic events, pulmonary embolism or other serious thromboembolic events; has major vascular diseases such as aortic aneurysm, aortic dissection aneurysm or other diseases that may endanger life or require surgery within 6 months prior to study intervention.
5. Uncontrolled systemic disease as judged by the investigator, included uncontrolled hypertension, uncontrolled diabetes, pesence of pleural effusion, pericardial effusion, or ascites that is clinically symptomatic or requires repeated drainage.
6. Patients with (noninfectious) interstitial lung disease (ILD) or history of pneumonia requiring steroid therapy; patients with serious pulmonary function impairment due to lung disease;
7. Patients with severe and/or uncontrolled concomitant diseases, such as decompensated cirrhosis of the liver, nephrotic syndrome, uncontrolled metabolic disorders, active inflammatory bowel disease or gastrointestinal perforation.
8. The toxicity from previous anti-tumor treatments has not yet recovered to ≤ grade 1 (based on the assessment of NCI CTCAE v5.0) or reached the level specified by the inclusion and exclusion criteria (excluding toxicities such as alopecia and fatigue that are judged by the investigators to be of low safety risk).
9. Has active autoimmune disease that has required systemic treatment in the past 2 years. Replacement therapy (eg, thyroxine, insulin, or physiologic corticosteroid) is allowed
10. Has diagnosis of immunodeficiency or is receiving chronic systemic steroid therapy (in dosing exceeding 10 mg daily of prednisone equivalent)
11. Known active tuberculosis;
12. Known history of allogeneic organ transplantation and allogeneic hematopoietic stem cell transplantation.
13. Certain viral infections including active hepatitis B or hepatitis C;
14. Known history of positive human immunodeficiency virus (HIV) test or known acquired immunodeficiency syndrome (AIDS); or positive syphilis antibody test;
15. Known hypersensitivity to the study drug or any of its components, or severe allergic reactions to other monoclonal antibodies;
16. Received any investigational anti-tumor vaccines or any drugs targeting the T-cell co-stimulation pathway;
17. Underwent major surgery within 20 days before study (as defined by the investigators) or were still in the recovery period of the previous surgery;
18. Has active infection requiring systemic therapy within 2 weeks
19. Received anticancer therapy in the adjuvant phase including but not limited to chemotherapy, small molecule tyrosine kinase inhibitors (TKIs), anti-tumor hormone therapy (except for LHRH agonists for mCRPC), systemic immunostimulants (including but not limited to interferons, IL-2), or approved anti-tumor indications of traditional Chinese medicine.
20. Pregnant or lactating women;
21. Local or systemic diseases caused by non-malignant tumors, or diseases or symptoms secondary to tumors, which may lead to higher medical risks and/or uncertainty in survival period evaluation, such as tumor leukemia-like reaction, cachexia manifestations, etc.
22. History of documented severe dry eye syndrome, severe Meibomian gland disease and/or blepharitis, or corneal disease that prevents/delays corneal healing

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 55 (Estimated)
Dates: Start 2025-08-01 (Estimated); Primary Completion 2027-12-31 (Estimated); Study Completion 2028-12-31 (Estimated)

PRIMARY OUTCOMES:
Objective Response Rate (ORR) | From baseline until disease progression, death or other protocol defined reason up to approximately 12 months
  ORR is defined as the proportion of subjects with confirmed CR or PR as the best overall response assessed per RECIST 1.1.
Adverse events (AEs) | From subject sign the ICF to 30 days after the last dose of study treatment
  Incidence and severity of adverse events (AEs) graded by Common Terminology Criteria for Adverse Events (CTCAE) v5.0.

CONTACTS AND LOCATIONS:
Overall Officials: Minghua Ge, Principal Investigator — Zhejiang Provincial People's Hospital